CLINICAL TRIAL: NCT05411211
Title: An Open-label, Multi-center, Post-marketing, Observational Study to Assess the Effectiveness and Safety of Adalimumab (Humira®) in Pediatric Patients With Polyarticular Juvenile Idiopathic Arthritis (pJIA) in China
Brief Title: An Observational Study to Assess Change in Disease Activity and Adverse Events of Adalimumab in Chinese Pediatric Participants With Polyarticular Juvenile Idiopathic Arthritis (pJIA)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-379
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Polyarticular Juvenile Idiopathic Arthritis
Keywords: Polyarticular juvenile idiopathic arthritis; pJIA; adalimumab; Humira
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric Participants receiving adalimumab: Pediatric Participants receiving adalimumab for polyarticular juvenile idiopathic arthritis (pJIA)

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common rheumatic disease affecting children, characterized by chronic synovitis with systemic multi-organ damage. Polyarticular juvenile idiopathic arthritis (pJIA) is a subtype of JIA defined as disease involving more than five joints in the first 6 months of disease. This study will assess how safe and effective adalimumab (Humira®) is in treating pediatric participants with pJIA in China real-world setting.

Adalimumab is an approved drug for the treatment of pJIA. Approximately 50 participants age 2 to 17 who are prescribed adalimumab for the treatment of pJIA in routine clinical practice will be enrolled at multiple sites in China.

Participants will receive adalimumab per their physician's usual prescription. Individual data will be collected for 52 weeks.

No additional study-related tests will be conducted during the routine physician visits. Only data which are routinely collected during a regular visit will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 2-17 years old with body weight ≥ 10kg.
* Diagnosis of polyarticular pJIA by treating physician.
* Adalimumab (Humira®) treatment is indicated as per Chinese label and according to judgement of the physician to Chinese clinical practice guidelines for the diagnosis and treatment of juvenile idiopathic arthritis.
* Participants or their parents/legal guardians are able and willing to give assent as well as informed consent approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) if applicable according to local law, and to comply with the requirements of this study protocol and Adalimumab (Humira ®) label.

Exclusion Criteria:

* Participants who cannot be treated with adalimumab according to Chinese Humira® label and by judgement of treating physician.
* Participants who receive any biological disease-modifying anti-rheumatic drugs (bDMARDs) within 6 months prior to the screening visit or who are on concomitant use of any bDMARD.
* Post menarche adolescent female subjects who are pregnant or breastfeeding or considering becoming pregnant during the study
* Participant is considered by the investigator or sub-investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Chinese Pediatric Participants with Polyarticular juvenile idiopathic arthritis (pJIA)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Physician's Global Assessment (PhGA) of Participant's Disease Activity by Visual Analog Scale (VAS) | Up to 52 Weeks
  PhGA measured by 100 mm VAS. VAS scores range from 0 to 100 points, 0=very good and 100=very bad.
Change from Baseline in Participants Experiencing Joint Pain | Up to 52 Weeks
  Participants Experiencing Joint Pain
Change from Baseline in Participants Experiencing Joint Swelling | Up to 52 Weeks
  Participants Experiencing Joint Swelling
Number of Active Joints Count | Up to 52 Weeks
  Active joints are defined as joints with swelling not due to deformity or joints with limitation of passive motion [LOM] and with pain and/or tenderness. Higher scores represent higher disease activity.
Number of joints with limitation of passive motion (LOM) | Up to 52 Weeks
  Number of joints with LOM
Number of joints with pain on passive motion (POM) | Up to 52 Weeks
  Number of joints with POM
Change from Baseline of C-Reactive Protein (CRP) and/or Erythrocyte Sedimentation Rate (ESR) levels | Up to 52 Weeks
  CRP and/or ESR level assessed as part of the physician's site routine car
Change from Baseline in Parent's or Child's Global Assessment of Participant's Disease Activity (Pa/ChGA) by Visual Analog Scale (VAS) | Up to 52 Weeks
  Pa/ChGA measured by 100 mm VAS. VAS scores range from 0 to 100 points, 0=very good and 100=very bad.
Change from Baseline in Physical function measured by Childhood Health Assessment Questionnaire (CHAQ) | Up to 52 Weeks
  The CHAQ assessed physical function. Scores go from 0= no disability to 3 = severe disability.
Change from baseline in dosage of corticosteroid | Up to 52 Weeks
Number of Participants with Adverse Events | Up to 52 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- China (2):
  - The Children's Hospital of Chongqing Medical University /ID# 232114, Chongqing, Chongqing Municipality
  - Wuhan Children's Hospital /ID# 242274, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-379#additional-resources-section